CLINICAL TRIAL: NCT03995771
Title: Adolescent Knee Pain (AK-Pain) Prognostic Tool
Status: Completed | Type: Observational
Sponsor: Aalborg University (Other)
Collaborators: TrygFonden, Denmark (Industry)
Responsible Party: Principal Investigator, Alessandro Andreucci, Dr. Alessandro Andreucci, post-doc researcher, Aalborg University
Other Study IDs: AAndreucci
Record Dates: First submitted 2019-06-15; First posted 2019-06-24 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Knee Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children and adolescents with knee pain: Children and adolescents (8-19 years old) presenting to general practice for knee pain
  Interventions: Other: Questionnaire delivery

INTERVENTIONS:
Other: Questionnaire delivery — A questionnaire including questions regarding prognostic factors for knee pain will be delivered to children and adolescents (8-19 years old) presenting to general practice with knee pain

SUMMARY:
The overall aim of this study is to develop and test a prognostic tool for knee pain in children and adolescents to be used in general practice.

By using the tool, general practitioners will be able to allocate the patient to a category of risk (e.g. low/medium/high) of recurrent or persistent knee pain at 3 months and 6 months, and to subsequently provide a treatment that is specific to the category of risk of the patient.

DETAILED DESCRIPTION:
One in three children and adolescents experience knee pain, and one in two will have a poor long-term prognosis with low quality of life and impaired physical activity levels.

Every year 119 - 200 children and adolescents per 10,000 registered patients consult their general practitioner for knee pain, and a variety of treatments are delivered, despite similar symptoms and patients' characteristics. However, the proportion of children and adolescents with a poor prognosis is high, which suggests that there is an urgent need to support the general practitioners in identifying those at high risk of a poor outcome early on, in order to better allocate resources.

This project will develop a user-friendly prognostic tool to support general practitioners' management of children and adolescents' knee pain.

Clinically relevant prognostic factors for child and adolescent knee pain were identified using systematic reviews and meta-analysis of individual participant data. Following feedback from general practitioners and children and adolescents on the content and understanding, the tool was piloted and implemented in general practice.

A cohort of approximately 300 children and adolescents will be recruited from general practices and followed-up for up to 6 months (the baseline starting date is July 2019 and the follow-up will end in July 2020) Clinically meaningful risk groups (e.g. low/medium/high) for the recurrence and persistence of knee pain (at 3- and 6-months) will be identified.

This tool will allow general practitioners to provide children and adolescents an optimal stratified care, by matching treatments to patients' prognostic profile.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents (aged 8-19 years old) who consult their general practitioner because of their knee pain (of both traumatic and non-traumatic origin) during a period of recruitment of 6 months (starting in July 2019)

Exclusion Criteria:

* Age below 8 years old or over 19 years old
* Consultation for musculoskeletal pain only in a body region different from the knee
* Pain originated by different conditions (e.g. cancer, infections)
* Child is vulnerable (e.g. he/she has experienced a recent trauma and the distress may have an impact on the self-report making it not valid)
* Inability to take part to the study because of inability to understand or comply

Ages: 8 Years to 19 Years | Sex: All
Age Groups: Child, Adult
Study Population: Children and adolescents (aged 8-19 years old) who consult their general practitioner because of their knee pain
Sampling Method: Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Recurrence/persistence of activity-limiting knee pain (i.e. yes/no pain that is limiting activities in the same knee) at 3-month follow-up | 3-month follow-up
  Activity-limiting knee pain: pain that is limiting activities in the same knee. Participants will also be asked about continuity of their knee pain (i.e. "how long have you been free of knee pain?"), to enable the distinction between recurrence (on/off knee pain episodes between baseline and follow-up) and persistence (continuous knee pain from baseline to follow-up) of knee pain

SECONDARY OUTCOMES:
Recurrence/persistence of activity-limiting knee pain (i.e. yes/no pain that is limiting activities in the same knee) at 6-month follow-up | 6-month follow-up
  Activity-limiting knee pain: pain that is limiting activities in the same knee. Participants will also be asked about continuity of their knee pain (i.e. "how long have you been free of knee pain?"), to enable the distinction between recurrence (on/off knee pain episodes between baseline and follow-up) and persistence (continuous knee pain from baseline to follow-up) of knee pain

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Andreucci, PhD, Principal Investigator — Aalborg University
Locations (1):
- Aalborg, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
A procedure is being developed for making data available to interested investigators.
  Investigators interested in using the data will have to apply through a data request procedure.
  Data access requests will be reviewed by a panel composed by the researchers participating to the project.
  Upon acceptance of the data request, a data access agreement will have to be signed.

REFERENCES:
- [Derived] Andreucci A, Holden S, Bach Jensen M, Skovdal Rathleff M. The Adolescent Knee Pain (AK-Pain) prognostic tool: protocol for a prospective cohort study. F1000Res. 2019 Dec 30;8:2148. doi: 10.12688/f1000research.21740.2. eCollection 2019. PMID 32399187
- See also: Webpage of the Center for General Practice at Aalborg University — http://www.generalpractice.aau.dk

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-15): https://cdn.clinicaltrials.gov/large-docs/71/NCT03995771/Prot_SAP_000.pdf